CLINICAL TRIAL: NCT04727359
Title: [Wissenschaftliche Evaluation Modellvorhaben in Der Kinder- Und Jugendpsychiatrie (§ 64b SGB V) - Therapeutische Intensivbehandlung im Ambulanten Setting (TIBAS) am Universitätsklinikum Tübingen]
Brief Title: Evaluation of a Flexible and Integrative Psychiatric Care Model in Child and Adolescent Psychiatry
Acronym: EVA_TIBAS
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Institute of Social Medicine and Health Systems Research, Medical Faculty, University Hospital Magdeburg (Unknown); Scientific Institut for Health Economics and Health System Research (WIG2) (Unknown)
Responsible Party: Principal Investigator, Anne Neumann, Principle Investigator, Technische Universität Dresden
Other Study IDs: EVA_TIBAS_01
Record Dates: First submitted 2021-01-15; First posted 2021-01-27 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Care; Cross-sectoral Treatment; Flexible and Integrated Treatment; FIT64b; Child and Adolescent Psychiatry; Evaluation; Cohort Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- FIT64b model project: Patients being treated in FIT64b model project at UKT
  Interventions: Other: FIT64b model project
- Standard care: Patients being treated in standard care (control hospitals)

INTERVENTIONS:
Other: FIT64b model project — FIT64b model project: The SHI funds AOK Baden-Württemberg and SVLFG (as an agricultural health insurance fund) have established a contract (duration = at least eight year) with the model hospital for an alternative remuneration / financing of patients treated in the model hospital (FIT64b hospital, UKT). This contract encourages the model hospital an alternative treatment of their patients (with the above mentioned SHI fund), for example fewer inpatient and more outpatient treatment.
  Groups: FIT64b model project

SUMMARY:
This study is an evaluation of the flexible and integrative psychiatric care model (according to § 64b of the German Social Code Book V (SGB V)) (FIT64b) in the child and adolescent psychiatry at the University Hospital Tübingen (UKT). The central concern of this evaluation is to answer the question whether FIT64b models offer advantages over standard care. The orientation of model care is a more cross-sectoral provision of services through more flexible treatment intensities.

DETAILED DESCRIPTION:
The introduction of Section 64b of the German Social Code, Book V (SGB V) created the possibility of agreeing so-called FIT64b model projects for the further development of care for mentally ill people. The objective is to improve cross-sectoral care or optimize patient care. The statutory health insurance (SHI) funds AOK Baden-Württemberg and the SVLFG (as an agricultural health insurance fund) have developed a FIT64b model project in child and adolescent psychiatry (KJP) with the UKT, which will be tested for a total of eight years in the care region of Tübingen starting on 01 October 2017. The core of the model care is the Therapeutic Intensive Treatment in the Outpatient Setting (TIBAS, from the German abbreviation of "Therapeutische Intensivbehandlung im Ambulanten Setting").

The goal of this model care is to provide more cross-sectoral service delivery through more flexible treatment intensities. The creation of TIBAS as an intensive outpatient form of treatment is intended to enable earlier discharge from the full inpatient setting. Four TIBAS levels have been implemented, representing different treatment intensities and frequencies, which can be flexibly deployed according to patient needs. A person-centered case manager accompanies patients throughout the treatment period. If necessary, the patients, but especially the family members, are accompanied by the social service of the AOK Baden-Württemberg and supported with regard to stabilizing the overall care situation (psychosocial counseling and networking with other care structures, etc.). For patients fulfilling the diagnostic criteria for either anorexia nervosa or moderate depression, direct access to TIBAS is possible without prior hospitalization.

The aim of the evaluation is to examine the achievement of the objectives of the FIT64b model project on the basis of anonymized claims data and primary data to be collected and to assess the transferability of the care approach to standard care. The main goals of the model project are to shorten the duration of inpatient stays while intensifying outpatient forms of treatment, to reduce the cumulative psychiatric treatment duration and the emergency admission rate, to reduce the symptom burden, to accelerate the return to psychosocial living conditions and to increase the quality of life. Stabilization of the family's overall care situation will be used to sustain these improvements. Through qualitative research methods, the experiences with and the subjective benefit of the social service of the AOK Baden-Württemberg as well as the cooperation of this social service with the UKT will be examined in more detail. The costs of the FIT64b model care should not exceed those of the standard care or, at a maximum of the same costs, better results should be achieved with regard to the above-mentioned patient-related goals.

The effectiveness, costs, and cost-effectiveness of the FIT64b model hospital compared to standard care are examined. The study presented here is a controlled cohort study which utilizes claims data as well as primary data. It will employ quantitative analyses of anonymized SHI data (Module A), quantitative analyses of questionnaires (Module B), and qualitative analyses of semi-structured interviews and a focus group (Module C). The controlled design is based on the fact that information of patients from the intervention hospital, the UKT, is compared to information of comparable patients from structurally similar hospitals of child and adolescent psychiatry in the same federal state (Petzold et al, Gesundheitswesen 2019, 81(1):63-71).

ELIGIBILITY:
Inclusion Criteria:

Module A

* treatment in UKT or control hospital (both KJP) within recruitment phase
* being insured with AOK Baden-Württemberg

Module B

* at least 6 years of age
* written consent of the children and adolescents plus written consent of the custodians
* sufficient cognitive and linguistic ability to participate in the survey

Module C1 (semi-structured interviews)

* sufficient knowledge of German as well as cognitive and linguistic abilities to participate in the interviews
* written consent of the custodians to participate
* recommendation for the social service of AOK Baden-Württemberg

Module C2 (focus group discussion) • several months of experience in working with the social service of the AOK Baden-Württemberg or the employees of the UKT within the framework of the FIT64b model project at the UKT

Exclusion Criteria:

Module A

* less than one year follow-up data available

Module B

• acute danger to self or others

Module C1 (semi-structured interviews) • none

Module C2 (focus group discussion)

• little cooperation with employees of the respective other institution (UKT and social service, e.g. one-time participation in a case conference)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Module A: anonymized data of the SHI fund AOK Baden-Württemberg, all patients being treated at the UKT or a control hospital between 01 January 2018 and 31 December 2021, claims data up to 31 December 2022 enabling an individual follow-up period of at least 12 months;
  Module B: all recruited patients being treated within 18-months recruitment phase starting in spring 2021 (and their custodians (e.g. parents or legal guardians) and siblings), in UKT and recruited control hospitals;
  Module C: C1: Semi-structured interviews: recruited parents (or legal guardians) of patients being treated within 18-months recruitment phase starting in spring 2021, only UKT, with recommendation for social service of the AOK Baden-Württemberg; C2: Focus group discussion: employees of UKT and social service
Sampling Method: Non-Probability Sample
Enrollment: 1037 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Duration of inpatient psychiatric treatment | one year prior to recruitment compared to first to fourth year after recruitment
  Days with inpatient stays of each included patient will be marked within the patient-individual follow-up period. A billing matrix defining the type of charge and describing the count will be used to mark days with inpatient stays. Inpatient stays that range outside the patient-specific follow-up time will be censored. The proportion of patients with at least one inpatient stay will be presented. Furthermore, the days of inpatient stays per patient will be added, including the stay that led to inclusion in the evaluation. The classification into inpatient and day care is based on the corresponding charges. If inpatient and day care cases are billed on one day in one hospital, this day will be counted as an inpatient day. It will be analyzed how long patients were treated in hospitals (here only inpatient stays), summed over the entire observation period for each case (all patients). (Module A)
Health related quality of life | cross-sectional analysis at baseline and / compared with follow-up 24 months after baseline
  The quality of life for patients will be measured using the KIDSCREEN-27 and compared between IG and CG. (Module B)

SECONDARY OUTCOMES:
Duration of day care psychiatric treatment | one year prior to recruitment compared to first to fourth year after recruitment
  Days with day care stays of each included patient will be marked within the patient-individual follow-up period. A billing matrix defining the type of charge and describing the count will be used to mark days with day care stays. Day care stays that range outside the patient-specific follow-up time will be censored. The proportion of patients with at least one day care stay will be presented. Furthermore, the days of day care stays per patient will be added, including the stay that led to inclusion in the evaluation. The classification into inpatient and day care is based on the corresponding charges. If inpatient and day care cases are billed on one day in one hospital, this day will be counted as an inpatient day. It will be analyzed how long patients were treated in hospitals (here only day care stays), summed over the entire observation period for each case (all patients). (Module A)
Inpatient psychiatric length of stay | one year prior to recruitment compared to first to fourth year after recruitment
  This outcome is similar to Outcome 1 with the difference that here it will be analyzed how long patients were treated in hospitals (only inpatient treatment), summed up over the time in hospital (i.e. only patients with hospital stays). (Module A)
Day care psychiatric length of stay | one year prior to recruitment compared to first to fourth year after recruitment
  This outcome is similar to Outcome 3 with the difference that here it will be analyzed how long patients were treated in hospitals (only day care treatment), summed up over the time in hospital (i.e. only patients with hospital stays). (Module A)
Outpatient psychiatric treatment in the hospital | one year prior to recruitment compared to first to fourth year after recruitment
  The number of days with a contact in the TIBAS care or the psychiatric outpatients departments (PIA) in the IG and CG will be recorded and compared. Since from 01.10.2017 the PIA care in the model project was merged into the TIBAS care and no separate PIA care took place in the IG from that date, here the TIBAS care will be considered as (intensive) outpatient treatment in the hospital and compared with the PIA care of the standard care. The annual and cumulative number of PIA contacts will be determined on the basis of the PIA documentation. (Module A)
Inpatient hospital readmission | first year after first full inpatient psychiatric discharge after recruitment
  The proportion of persons with an inpatient stay who were readmitted as inpatients within one year after discharge from the hospital and the days between first inpatient discharge and second inpatient treatment will be examined. The follow-up period is determined on a patient-specific basis. For this purpose, the first discharge date from an inpatient stay in the reference hospital (IG or CG) after inclusion into the evaluation that allowed a one-year follow-up period will be taken as the basis. Readmission is given if the patient had a psychiatric diagnosis (ICD-10: Fx) as main diagnosis and was readmitted with a psychiatric diagnosis as main diagnosis within one year. (Module A)
Emergency admission rate | one year prior to recruitment compared to first to fourth year after recruitment
  The proportion of inpatient cases with admission reason xxx7 (emergency admission) will be extracted. The proportion of patients with a psychiatric diagnosis and emergency admission will be analyzed in relation to all inpatient admissions with a psychiatric diagnosis at the reference hospital. (Module A)
Direct medical care costs | one year prior to recruitment compared to first to fourth year after recruitment
  The difference in the costs for the treatment of mental illnesses arising between IG and CG during the observation period taking a SHI-funds perspective will be analyzed. In addition, somatic costs will be estimated. For this purpose, the care costs of the following areas will be taken into account: costs of inpatient and day care, costs of TIBAS care, cost of outpatient care in hospitals, costs of SHI-accredited medical care, drug costs and remedies costs. (Module A)
Cost-effectiveness (direct medical costs) | one year prior to recruitment compared to first to fourth year after recruitment
  To compare the efficiency of the model project with standard care, a cost-effectiveness analysis will be performed taking a SHI-funds perspective. The incremental cost-effectiveness ratio will be determined using the primary outcome parameter cumulative duration of inpatient stays as the effect measure. (Module A)
Symptom burden | cross-sectional analysis at baseline and / compared with follow-up 24 months after baseline
  The symptom burden will be measured using the Strengths and Difficulties Questionnaire (SDQ) and compared between IG and CG. (Module B)
Return to psychosocial relationships | cross-sectional analysis at baseline and / compared with follow-up 24 months after baseline
  The return to psychosocial relationships will be measured using a self-developed questionnaire covering areas of friends, school, sports activities, hobbies, social integration and daily structure and compared between IG and CG. (Module B)
Treatment satisfaction | cross-sectional analysis at baseline and / compared with follow-up 24 months after baseline
  Treatment satisfaction will be measured using the Treatment assessment questionnaire (FBB ("Fragebogen zur Beurteilung von Behandlungen")) and compared between IG and CG. (Module B)
Societal costs | cross-sectional analysis at baseline and / compared with follow-up 24 months after baseline
  The costs of the treatment due to mental illnesses from a societal perspective will be estimated using an adapted questionnaire based on the Client Sociodemographic and Service Receipt Inventory (CSSRI) questionnaire. (Module B)
Cost-effectiveness (societal costs) | cross-sectional analysis at baseline and / compared with follow-up 24 months after baseline
  Cost-effectiveness will be estimated comparing the results from the quality of life and the societal costs comparing IG and CG. (Module B)
Offer and effects of social service (qualitative data) | cross-sectional, semi-structured interviews conducted between spring 2021 and summer 2022
  Semi-structured interviews with families using a self-developed interview guide with open-ended questions will be used. (Module C)
Benefit social service (qualitative data) | cross-sectional, semi-structured interviews conducted between spring 2021 and summer 2022
  Semi-structured interviews with families using a self-developed interview guide with open-ended questions will be used. (Module C)
Cooperation (strengths and potentials for optimization) between UKT and social service employees (qualitative data) | cross-sectional, focus group discussion conducted between spring 2021 and summer 2022
  Self-developed open-ended questions in a focus group discussion will be used. (Module C)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Neumann, PhD, Principal Investigator — Technische Universität Dresden
Locations (1):
- Universitätsklinikum Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petzold T, Neumann A, Seifert M, Kuster D, Pfennig A, Weiss J, Hackl D, Swart E, Schmitt J. [Identification of Control Hospitals for the Implementation of the Nationwide and Standardized Evaluation of Model Projects According to section sign 64b SGB V: Analysis of Data from Structured Quality Reports]. Gesundheitswesen. 2019 Jan;81(1):63-71. doi: 10.1055/s-0042-116436. Epub 2016 Nov 15. German. PMID 27846670
- [Derived] Neumann A, Hense H, Baum F, Kliemt R, Seifert M, Harst L, Kubat D, Maicher B, Schrey C, Schmitt J, Pfennig A, Weinhold I, Swart E, Soltmann B. Evaluation of a flexible and integrative psychiatric care model in a department of child and adolescent psychiatry in Tubingen, Germany: study protocol (EVA_TIBAS). BMC Health Serv Res. 2021 Nov 22;21(1):1262. doi: 10.1186/s12913-021-07226-1. PMID 34802427